CLINICAL TRIAL: NCT06052189
Title: Use of Ultrasonographic Parameters in Preoperative Prediction of Difficult Laryngoscopy in Non-suspected Difficult Airway Patients Undergoing Elective Surgery; a Prospective Observational Study
Brief Title: Ultrasonographic Parameters in Prediction of Difficult Laryngoscopy in Non-suspected Difficult Airway Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Eldein Shalaby Abotaleb, Resident of Anesthesiology, Surgical ICU, and Pain therapy, Tanta University
Other Study IDs: 35566/6/22
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Ultrasound; Difficult Laryngoscopy; Prediction
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Easy laryngoscopy: Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.
  Interventions: Procedure: Ultrasound
- Difficult laryngoscopy: Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasonographic parameters: in the parasagittal plane (1cm from midline) with the patient lying supine, without a pillow, head, and neck in the neutral position, looking straight ahead with mouth closed and the tongue on the floor of the mouth without any movement.

SUMMARY:
This study aims to evaluate the ultrasonographic parameters (distance from skin to epiglottis (DSE) and distance from skin to vocal cords (DSVC)) as preoperative predictors of difficult laryngoscopy in non-suspected difficult airway patients undergoing elective surgery.

DETAILED DESCRIPTION:
Airway management is an integral part of general anesthesia. It simply aims to secure the patient's airway and achieve adequate ventilation and oxygenation for the patient undergoing surgery under general anesthesia. Unsuccessful airway management due to the unexpected difficulty in laryngoscopy is a life-threatening situation and may lead to morbidity and mortality.

Many conventional clinical tests are used in preoperative airway assessment such as modified Mallampati classification, Thyro-mental distance, inter-incisor distance, cervical mobility, and neck circumference, which are used to predict difficulty in the airway, but they have limited value and low sensitivity and specificity. Difficult laryngoscopy cannot be always predicted based on the preoperative assessment by conventional clinical tests. Some patients are thought to have an easy airway by clinical tests, but they show an unexpected difficulty in the laryngoscopy.

The laryngeal view of the patient can be assessed and graded during direct laryngoscopy using the Cormack and Lehane grading scale and its modification that describes the laryngoscopy as easy or difficult.

Ultrasonography is a valuable promising tool for preoperative airway evaluation through identifying important sonoanatomy of the upper airway such as epiglottis, thyroid cartilage, and vocal cords.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 65 years.
* Both sexes.
* Patients who aren't suspected to have a difficult airway after preoperative airway assessment by conventional clinical tests such as modified Mallampati classification (MMC), thyromental distance (TMD), inter-incisor distance (IID), cervical mobility (CM), And neck circumference (NC).
* American society of anesthesia (ASA) I, II, and III physical status.
* Scheduled for elective surgery under general anaethesia.

Exclusion Criteria:

* Patients with maxillofacial injury and airway trauma.
* Patients with a history of previous difficult intubation.
* Patients with anatomical abnormalities.
* Neck scarring, swelling, or burn.
* Pregnancy.
* Obesity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective observational study will be carried out on 85 patients at Tanta University Hospital in the anesthesia department over a period of one year from May 2022 to May 2023, which may be extended after approval from the institutional ethical committee of the faculty of medicine at Tanta University.
  Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Correlation between the ultrasonographic parameters and the modified Cormack and Lehane grading scale | 10 minutes during intubation.
  Correlation between the ultrasonographic parameters (distance from skin to epiglottis ( DSE) and distance from skin to vocal cords (DSVC)) and the modified Cormack and Lehane grading scale of laryngoscopy as easy or difficult

SECONDARY OUTCOMES:
Sensitivity of ultrasonographic distance from skin to epiglottis to predict difficult laryngoscopy. | 10 minutes during intubation.
  Measurement of Sensitivity of ultrasonographic distance from skin to epiglottis to predict difficult laryngoscopy.
  Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.
Sensitivity of ultrasonographic distance from skin to vocal cords to easy laryngoscopy. | 10 minutes during intubation.
  Measurement of Sensitivity of ultrasonographic distance from skin to epiglottis to predict easy laryngoscopy.
  Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.
Specificity of ultrasonographic distance from skin to epiglottis to predict difficult laryngoscopy. | 10 minutes during intubation.
  Measurement of Specificity of ultrasonographic distance from skin to epiglottis to predict difficult laryngoscopy.
  Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.
Specificity of ultrasonographic distance from skin to vocal cords to easy laryngoscopy. | 10 minutes during intubation.
  Measurement of Specificity of ultrasonographic distance from skin to epiglottis to predict easy laryngoscopy.
  Laryngeal view grading according to the modified Cormack and Lehane grading scale where grades 1 and 2a are considered easy laryngoscopy and grades 2b, 3, and 4 are considered difficult laryngoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of the study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of the study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.